CLINICAL TRIAL: NCT07236021
Title: Promoting Emotion Regulation in Patients Living With Chronic Cancer : A Pilot Feasibility, Acceptability and Tolerability Study (e-Motion Project)
Brief Title: e-Motion : Promoting Emotion Regulation in Chronic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: Centre de Psycho-Oncologie (CPO) (Other); Jules Bordet Institute (Other); Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Isabelle Merckaert, Professor, Université Libre de Bruxelles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PO20250132
Record Dates: First submitted 2025-09-05; First posted 2025-11-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Cancers; Myeloma Multiple
Keywords: Advanced cancer; Cognitive Behavioral Therapy (CBT); Emotional regulation; Ecological Momentary Assessment (EMA); Hypnosis; Psychotherapy Group
MeSH Terms: conditions — Neoplasms; Multiple Myeloma; Emotional Regulation | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: A pilot feasibility, acceptability and tolerability project. Two steps: The first included 15 patients will be assigned to a Guided Self-Help intervention. The second starts only after the first has ended. For this one, 15 other patients are recruited and assigned to a Group and Guided Self-Help intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Self-Help intervention arm (Active Comparator): Guided self-help emotion regulation intervention for patient with chronic and incurable cancer.
  Interventions: Behavioral: Guided Self-Help intervention
- Group and Guided Self-Help intervention arm (Experimental): Group and guided self-help emotion regulation intervention for patient with chronic and incurable cancer.
  Interventions: Behavioral: Group and Guided Self-Help intervention

INTERVENTIONS:
Behavioral: Guided Self-Help intervention — This intervention will consist of 8 self-administered modules that patients will complete every week.
  The sessions integrate an emotion regulation component with breathing exercises, relaxation exercises, hypnosis, etc. Once a week (maximum 15-minute), a trained psychologist will call the patient to help and/or encourage them. Each module will consist of podcasts, a reading assignment (with psycho-educational information) and writing assignments. The intervention will include home exercises and patients will be encouraged to practice exercises and skills learned between the sessions.
  Arms: Guided Self-Help intervention arm
Behavioral: Group and Guided Self-Help intervention — It will consist of the same content described above, but given in 8 group sessions (2-hour) held by videoconference (Zoom) that will take place every week. Patients will also have access to the podcasts, home exercises and reading assignment, but will benefit from increased motivation and support from both the therapist and their peers in the group. Each group will be composed of 5 patients.
  Arms: Group and Guided Self-Help intervention arm

SUMMARY:
The present study aimed to pilot evaluate two interventions: a Guided Self-Help Intervention alone, and a combined Group and Guided Self-Help Intervention, designed to support individuals living with chronic cancer and recently diagnosed. The primary aim of this pilot study is to assess the feasibility, acceptability and tolerability of the interventions. The secondary aim of the pilot study is to assess the interventions preliminary efficacy and differences on psychological symptoms.

DETAILED DESCRIPTION:
The investigators aim to conduct a pilot study to assess feasibility, acceptability and tolerability of two interventions on 30 chronic cancer patients: a Guided Self-Help Intervention and a combined Group and Guided Self-Help Intervention. Both interventions will rely on emotion regulation component, with CBT, hypnosis, and positive psychology techniques.

The first 15 patients that will be recruited will be allocated to the Guided Self-Help Intervention (Arm 1). The recruitment of the 15 other patients will start after the last assessment of the last patient included in the first arm. These 15 other patients will be allocated by group of 5 to the combined Group and Guided Self-Help Intervention (Arm 2). Each participants will be assessed before intervention (T1), during intervention (Ecological weekly assessment, week 1 to week 12) and after the intervention (T2, 15 weeks after T1). T1 and T2 assessments will include self-reported questionnaires about psychological symptoms and a 7-day ecological momentary assessment (EMA) on emotions. In T2, a semi-structured interview will be performed for each participant to collect qualitative information on the tolerability and acceptability of the interventions. Participants will also complete a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Having received a diagnosis of chronic cancer (metastatic breast cancer, metastatic melanoma, metastatic colorectal, metastatic ovarian, metastatic uterine, metastatic endometrial, metastatic prostate, metastatic bladder, metastatic kidney or metastatic testicular cancer, symptomatic multiple myeloma, metastatic non-small cell lung, metastatic mesothelioma or metastatic thymoma) in the past 12 months,
* Having completed at least one active treatment session (e.g., chemotherapy, surgery, radiotherapy, immunotherapy, target therapy).

Exclusion Criteria:

* Having less than one year of life expectancy
* Having more than one treatment line (for triple negative breast cancer, melanoma, gynecological cancer, colorectal cancer, bladder cancer, kidney cancer, non-small cell lung, mesothelioma and thymoma) or two treatment lines (for other breast cancers and testicular cancer) or three treatment lines (for prostate cancer and multiple myeloma),
* Having a diagnosis of oligometastatic cancer,
* Age < 18 years,
* Non-fluency in French,
* Inability to follow the online intervention,
* Severe cognitive impairment, and severe and/or acute psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline (T0)
  At least 25% of eligible patients agree to participate.
Retention rate | Baseline (T0), Weekly 15 (T2)
  At least 80% of patients complete the study to the end. The study completion rate is calculated based on the difference between the number of patients enrolled in T0 and those who completed the study in T2.
Adherence to intervention | Weeks 1 to 12 (intervention with weekly call)
  At least 70% of patients complete all sessions regardless of the intervention arm. The weekly call includes a question asking participants whether they attended the week's session. Answer with Yes or No. If yes: go through all of the following questions. If no: investigate further to see if anything has been done."
Adherence to between-session practice | Weeks 1 to 12 (intervention with weekly call)
  At least 70% of patients complete all assigned between-session exercises. The weekly call includes a question asking participants if they have done their exercises throughout the week. Answer with yes or no. The exercise completion rate between sessions is defined as the proportion of patients who reported having completed all weekly exercises among those who responded to the follow-up question.
Data completeness self-report questionnaire | Baseline (T1) and Weekly 15 (T2)
  At least 90% of patients complete all data of questionnaires at both time points (T1 and T2).
Data completeness EMA | Baseline (T1), Weeks 1 to 12 (Ecological weekly assessment), Weekly 15 (T2)
  At least 70% of data are collected for the ecological momentary assessments.
Satisfaction of the intervention | Week 15 (T2)
  At least 80% of patients rate the intervention as satisfactory. This percentage is calculated based on the response to one of the questions in the satisfaction questionnaire, which is 1-item, 6-point self-report questionnaire (0 = Not at all, 6 = Absolutely). The question investigates whether, overall, participants were satisfied with the intervention. Mean score is ≥ 4 in the satisfaction questionnaire. Satisfaction will also be assessed through a qualitative analysis (thematic analysis) of the transcript of the exit interview. The questionnaires were developed for this study.
Willingness to recommend | Week 15 (T2)
  At least 80% of patients would recommend the intervention to other patients. This percentage is calculated based on the response to one of the questions in the satisfaction questionnaire, which is 1-item, 6-point self-report questionnaire (0 = Not at all, 6 = Absolutely). The question investigates the extent to which participants would recommend this intervention to other patients in their situation. Mean score is ≥ 4 in the satisfaction questionnaire. The questionnaire was developed for this study.
Dropout rate due to intervention-related burden | Baseline (T1), Weeks 1 to 12 (Intervention), Weekly 15 (T2)
  No more than 10% of patients discontinue participation due to emotional distress or perceived burden linked to the intervention, as assessed by one question of the drop-out questionnaire which is: 'The reasons for this decision are related to: A. The intervention B. The questionnaires C. Both.' The percentage is calculated based on the number of patients who answered A or C.
Self-reported emotional impact | Week 15 (T2)
  At least 80% of patients indicate that the intervention was emotionally manageable and not overly distressing. This percentage is calculated based on the response to one of the questions in the satisfaction questionnaire, which is 1-item, 6-point self-report questionnaire (0 = Not at all, 6 = Absolutely). The question investigates the extent to which participants found this intervention emotionally comfortable or bearable. Mean score is ≥ 4 in the satisfaction questionnaire. Self-reported emotion impact will also be based on responses from the exit interviews (which is a semi-structured interview), assessed through a qualitative analysis (thematic analysis). The questionnaires were developed for this study.

SECONDARY OUTCOMES:
The Generalized Anxiety Disorders 7 items (GAD-7) | Baseline (T1), Week 15 (T2)
  The preliminary efficacy and interventions differences will be assessed using self-report questionnaires. The GAD-7, which is a validated 7-item, 4-point self-report questionnaire assessing anxiety symptoms. A higher score indicates higher levels of anxiety.
The Patient Health Questionnaire 9 items (PHQ-9) | Baseline (T1), Week 15 (T2)
  The preliminary efficacy and interventions differences will be assessed using self-report questionnaires. The PHQ-9 which is a validated 10-item, 4-point self-report questionnaire assessing depressive symptoms. A higher score indicates higher levels of depression.
The Penn State Worry Questionnaire (PSWQ) | Baseline (T1), Week 15 (T2)
  The preliminary efficacy and interventions differences will be assessed using self-report questionnaires. The PSWQ which is a validated 16-item, 5-point self-report questionnaire assessing worry. A higher score indicates higher levels of worry.
Fear of Cancer Recurrence Inventory (FCRI) | Baseline (T1), Week 15 (T2)
  The preliminary efficacy and interventions differences will be assessed using self-report questionnaires. The FCRI (Fear of cancer progression modified Fear of Cancer Recurrence Inventory) : which is a validated 42-item, 5-point self-report questionnaire assessing seven dimensions of fear of cancer recurrence (0 = Never, 4 = All the time): triggers, severity, psychological distress, coping strategies, functioning impairments, insight, and reassurance. This scale has been validated in patients with metastatic cancer. However, to simplify the understanding of the items, the investigators have adapted it by substituting "fear of cancer recurrence" by "fear of cancer progression". Higher score indicates higher levels of fear of cancer progression.
Self-efficacy | Baseline (T1), Week 15 (T2)
  The preliminary efficacy and interventions differences will be assessed using self-report questionnaires. The self-efficacy questionnaire was designed to assess patients' confidence in their ability to effectively manage and regulate their emotions. Self-efficacy was assessed using a questionnaire developed for this study, which is a 13 items on a 10-point Likert scale (0 = Not at all certain, 10 = Absolutely certain).

CONTACTS AND LOCATIONS:
Overall Officials: Florence Lewis, PhD, Principal Investigator — Université Libre de Bruxelles; Isabelle Merckaert, Professor, Study Director — Université Libre de Bruxelles
Locations (2):
- Belgium (2):
  - Institut Jules Bordet, Hôpital universitaire de Bruxelles, Brussels, Anderlecht
  - H.U.B Institut Jules Bordet, Brussels, Brussels Capital

IPD SHARING:
Plan to Share IPD: No